CLINICAL TRIAL: NCT06960122
Title: Clinical Study on Fecal Microbiota Transplantation for Diarrhea After Total Pancreatectomy
Acronym: FMT-TP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Principal Investigator, caiwen, Chief Physician, Second Affiliated Hospital, School of Medicine, Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-0303
Record Dates: First submitted 2025-04-10; First posted 2025-05-07 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-04

CONDITIONS: Pancreatic Cancer, Resected; Diarrhea
MeSH Terms: conditions — Pancreatic Neoplasms; Diarrhea | interventions — Fecal Microbiota Transplantation; Standard of Care

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fecal microbiota transplantation (Experimental): One course of fecal microbiota transplantation (FMT) was administered in addition to standard therapy.
  Interventions: Procedure: Fecal Microbiota Transplant (FMT)
- Control (Active Comparator): Standard Therapy Alone
  Interventions: Other: Standard Therapy

INTERVENTIONS:
Procedure: Fecal Microbiota Transplant (FMT) — One course of fecal microbiota transplantation (FMT) was administered in addition to standard therapy.
  Arms: Fecal microbiota transplantation
Other: Standard Therapy — Standard Therapy Alone
  Arms: Control

SUMMARY:
By 2030, pancreatic cancer is projected to become the second leading cause of cancer-related deaths, with a 5-year survival rate below 10%. Approximately 20% of patients are diagnosed at a borderline resectable or resectable stage, and surgical resection remains the only curative option. However, total pancreatectomy (TP) often leads to severe diarrhea (incidence rate: 43.5%) due to exocrine insufficiency, and current pancreatic enzyme replacement therapy shows limited efficacy in some patients.

Recent studies highlight the critical role of gut microbiota in pancreatic cancer progression and postoperative recovery. Patients with pancreatic ductal adenocarcinoma (PDAC) exhibit a 1000-fold increase in intrapancreatic bacterial load compared to normal tissues, with significantly elevated Bacteroides abundance and reduced Firmicutes and Proteobacteria in fecal samples. Postoperative dysbiosis is linked to complications; for example, diarrhea after cholecystectomy is dominated by Proteobacteria, suggesting that microbial imbalance may underlie diarrhea following TP.

To address this, the study proposes fecal microbiota transplantation (FMT) via oral capsules. FMT has proven effective in treating recurrent Clostridium difficile infection by restoring healthy microbiota. This research will systematically evaluate the efficacy and safety of FMT in alleviating post-TP diarrhea through clinical indicators and 16S rDNA sequencing, offering novel insights into postoperative management of pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years, regardless of gender.
2. Anticipated survival ≥3 months.
3. Severe post-total pancreatectomy diarrhea (as per HART score).
4. Willing and able to provide written informed consent and complete follow-up assessments.
5. Eastern Cooperative Oncology Group (ECOG) performance status score of 1-3.
6. No use of oral/intravenous broad-spectrum antibiotics within 3 days prior to enrollment.
7. Ability to swallow capsules intact without chewing.
8. Adequate organ function confirmed by screening-phase laboratory tests.

Exclusion Criteria:

1. Major organ insufficiency/failure, including but not limited to:

   Cardiac insufficiency or heart failure Renal insufficiency or renal failure Hepatic insufficiency or liver failure
2. Uncontrolled or severe infections.
3. Documented history of:

   Psychoactive drug abuse Alcoholism Illicit drug use
4. Severe infections complicated by sepsis or septicemia.
5. History of severe allergic reactions or known hypersensitivity to components of liquid live-bacterial enteric-coated capsules.
6. Pregnancy or lactation, or women of childbearing potential refusing contraceptive measures during the 15-week observation period.
7. Gastrointestinal perforation and/or fistulas.
8. Other conditions deemed ineligible by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Diarrhea HART Score | Assessed every two cycles up to 24 weeks (each cycle is 21 days)
  The Hart Diarrhea Scoring Scale assigns scores to nine categories. The total score is the sum of scores from each bowel movement on the same day, with each movement evaluated using this scale. A cumulative score of ≥12 points within 24 hours is classified as diarrhea.

SECONDARY OUTCOMES:
Gastrointestinal Symptom Rating Scale (GSRS) | Assessed every two cycles up to 24 weeks (each cycle is 21 days)
  The total score of the GSRS (Gastrointestinal Symptom Rating Scale) ranges from 0 to 78 points, with higher scores indicating more severe gastrointestinal symptoms in patients.
Quality of Life (QoL) assessment | Assessed every two cycles up to 24 weeks (each cycle is 21 days)
  The maximum score is 60. A score of less than 20 indicates an extremely poor quality of life; 21-30, poor; 31-40, fair; 41-50, relatively good; and 51-60, good.
Chemotherapy cycle delay rate | Assessed every two cycles up to 24 weeks (each cycle is 21 days)
Colonization status of intestinal beneficial flora | At baseline, completion of 4 intervention cycles, and completion of 8 intervention cycles (each cycle is 21 days)
  Stool samples were collected from patients at three time points: baseline, after 4 cycles of intervention, and after 8 cycles of intervention, for 16S rDNA sequencing.

CONTACTS AND LOCATIONS:
Overall Officials: Wen Cai, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No